CLINICAL TRIAL: NCT07124455
Title: Investigation of Respiratory Muscle Strength, Endurance, and Postural Control in Individuals With Non-Specific Chronic Neck Pain and Varying Degrees of Disability
Brief Title: Respiratory Muscle Strength, Endurance, and Postural Control in Chronic Neck Pain With Disability
Acronym: ISU BT 1
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Beyza Tanrıöğen, Research Assistant (PhD student), Istinye University
Other Study IDs: IstinyeU BT 1
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Neck Pain Chronic; Respiratory Function
Keywords: neck pain; respiratory function; neck disability; respiratory muscle strength; pain
MeSH Terms: conditions — Respiratory Aspiration; Neck Pain; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy individuals: participants without neck pain
- mild: participant with mild neck disability according to neck disavility index
- moderate: participant with moderate neck disability according to neck disavility index
- severe: participant with severe neck disability according to neck disavility index

SUMMARY:
Neck pain is a common cause of disability worldwide, especially among middle-aged women in wealthy countries. It often occurs in episodes and can become chronic, affecting physical, psychological, emotional, and social aspects of life, which reduces quality of life for both patients and their families. Research has shown that neck pain is linked to problems with movement control, such as reduced neck mobility, increased activity in surface muscles, and poor body position awareness. These issues may lead to breathing problems because surface neck muscles are involved in inhalation. Studies have found that people with chronic neck pain have reduced lung function and altered breathing patterns compared to healthy individuals. However, no research has yet explored how respiratory endurance and balance control relate to neck pain severity. This study will assess respiratory muscle strength, endurance, and postural control in people with chronic neck pain. Participants will be divided into groups based on the severity of their neck disability, and their respiratory and balance measurements will be compared to healthy individuals. The goal is to understand whether worsening neck disability is associated with greater respiratory problems.

DETAILED DESCRIPTION:
This study designed as cross-sectional study. Aim

The aim of this study is to investigate the presence of respiratory dysfunction in individuals with chronic non-specific neck pain by evaluating respiratory muscle strength, endurance, and postural control. It also aims to classify the data obtained according to the severity of neck disability and to determine whether respiratory dysfunction is associated with the severity of neck involvement.

Research Hypotheses

H0: There is no difference in respiratory muscle strength, endurance, and postural control parameters between individuals with chronic non-specific neck pain and asymptomatic individuals.

H1: There is a difference in respiratory muscle strength, endurance, and postural control parameters between individuals with chronic non-specific neck pain and asymptomatic individuals.

H2: The severity of chronic non-specific neck pain has no effect on the degree of respiratory impairment.

H3: The severity of chronic non-specific neck pain has an effect on the degree of respiratory impairment.

Specific Objectives of the Study

To assess the severity of neck pain using the Neck Disability Index

To measure the respiratory muscle strength of participants

To measure the respiratory muscle endurance of participants

To evaluate the postural control of participants

To compare respiratory muscle strength, endurance, and postural control between individuals with neck pain and asymptomatic participants

To examine the relationship between the severity of neck pain and the extent of respiratory dysfunction

ELIGIBILITY:
Inclusion Criteria:

Individuals diagnosed with Non-Specific Neck Pain by a physician

Having complaints of Non-Specific Neck Pain for at least 3 months

Aged between 18 and 65 years

Willingness to participate voluntarily

No diagnosed respiratory disease

No diagnosed cardiac disease

No diagnosed neuromuscular disease

Non-smoker

Exclusion Criteria:

Presence of radiculopathy or structural abnormalities in the cervical region

History of surgery on the cervical region

Upper respiratory tract infection within the last 3 months

History of surgery involving the chest cage or spine

Spinal deformities such as scoliosis or kyphosis

History of abdominal surgery

Inflammatory and rheumatological diseases

Presence of infection in the bone or soft tissue of the cervical spine

Presence of malignancy

Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people with chronic non-specific neck pain
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
respiratory function test | 4 weeks
  Lung function will be measured with a portable spirometer. The test will record forced vital capacity, the amount of air exhaled in one second, their ratio, and peak flow. Results will be given in liters and compared to predicted normal values. The test follows official guidelines and uses sterilized, personal mouthpieces to ensure safety.
Maximum Inspiratory Pressure | 4 weeks
  Maximum inspiratory mouth pressure is the intraoral pressure measured during maximum inspiration against a closed airway valve. For the measurement, the participant is asked to perform a maximum expiration first. Then, the airway valve is closed, and the participant performs a maximum inspiration, maintaining it for 1-3 seconds. The best value out of three attempts will be selected and recorded in cmH₂O. Results will be expressed as a percentage of normal reference values calculated according to age and gender.
Assessment of Cervical Disability: | 4 weeks
  Cervical disability will be evaluated using the Turkish version of the Neck Disability Questionnaire. This is one of the most commonly used questionnaires for neck pain. It is used to assess the patient's current condition and progress during treatment. The questionnaire consists of 10 sections completed by the patient, covering pain, personal care, lifting heavy objects, reading, headaches, concentration, work, driving, sleeping, and recreation. Each section is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no disability) to 50 (total disability). An increase in the score indicates greater disability, while a decrease indicates improvement. Based on the total score, disability is classified as follows: 0-4 points (0-8%) no disability, 5-14 points (10-28%) mild disability, 15-24 points (30-48%) moderate disability, 25-34 points (50-64%) severe disability, and 35-40 points (70-100%) complete disability (Vernon et al., 1991; Telci et al., 2009).
Measurement of Respiratory Muscle Endurance | 4 weeks
  Respiratory muscle endurance refers to the ability of the respiratory muscles to sustain performance during prolonged or repetitive contractions. This parameter is typically assessed with specific endurance tests and may vary depending on the measurement protocol. During the endurance test, the participant sustains respiratory muscle activity under a given load or intensity for a specified duration, and performance values are recorded.
Maximum Expiratory Pressure | 4 weeks
  Maximum Expiratory Pressure is the intraoral pressure measured during maximum expiration against a closed airway valve. For the measurement, the participant first performs a maximum inspiration. Then, the airway valve is closed, and the participant performs maximum expiration, maintaining it for 1-3 seconds. The highest value out of three attempts will be selected and recorded in cmH₂O. Results will be expressed as a percentage of normal reference values calculated according to age and gender.

SECONDARY OUTCOMES:
Anthropometric Measurements: | 4 weeks
  Waist circumference and chest circumference measurements at three different regions will be taken.
Postural Analysis: | 4 weeks
  For postural analysis, the form developed by Corbin et al. will be used. Scoring will be performed according to the severity of postural deviations observed from the lateral and posterior views (Corbin et al., 2006).
Visual Analog Scale: | 4 weeks
  Perceived exertion, fatigue, and breathlessness will be assessed using the Visual Analog Scale (VAS) ranging from 0 (none) to 10 (very severe).
Assessment of Postural Control: | 4 weeks
  The Functional Reach Test will assess postural control using a tape fixed to a wall. Participants stand close to the wall and reach forward with their dominant arm without stepping or lifting heels. Three trials will be done, averaging the last two. Before testing, handedness will be determined. Modified tests include reaching with both arms and on soft surfaces, as well as reaching sideways.
Borg Scale: | 4 weeks
  Perceived exertion, fatigue, and breathlessness will be assessed using modified Borg scale, ranging from 0 (none) to 10 (very severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No